CLINICAL TRIAL: NCT03844204
Title: Effect of a Servo-control System on Heat Loss in Very Low Birth Weight Infants at Birth: a Multicenter, Prospective, Randomized Controlled Trial
Brief Title: Effect of a Servo-control System on Heat Loss in Very Low Birth Weight Infants at Birth
Acronym: SCOPRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Padova (Other)
Responsible Party: Principal Investigator, Daniele Trevisanuto, Professor, University Hospital Padova
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 4371/AO
Record Dates: First submitted 2019-02-14; First posted 2019-02-18 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Neonatal Hypothermia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Nurses who will measure the temperature at NICU admission are blind to treatment arm in the delivery room
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Servo-controlled system (Experimental): The temperature probe of the servo-controlled system will be positioned on the patient's abdomen with an adhesive tape. The body temperature will be set at 37°C.
  Interventions: Device: Thermal servo-controlled system
- No servo-controlled system (Active Comparator): The temperature of the infant warmer will be manually set at maximum of power output.
  Interventions: Device: Thermal servo-controlled system

INTERVENTIONS:
Device: Thermal servo-controlled system — All patients will be positioned under the infant warmer. In the treatment group, a probe positioned on the skin of the neonate will guide the thermal exposure in a servo-controlled modality. In the control group, thermal exposure will be determined manually by setting the power of the heater at the maximum output.

SUMMARY:
Hypothermia in preterm infants during the immediate postnatal phase is associated with morbidity and mortality and remains an unresolved, worldwide challenge.

A list of interventions, including adequate room temperature, use of infant warmers, polyethylene bags/wrap, pre-heated mattresses, caps and heated and humidified gases, to prevent thermal loss at birth in very preterm infants has been recommended, but a certain percentage of very preterm infants are hypothermic at the time of the neonatal intensive care unit (NICU) admission suggesting that further measures are needed. The thermal servo-controlled systems are routinely used in the NICU to accurately manage the patients' temperature, but their role during the immediate postnatal phase has not been previously assessed.

We hypothesized that using a thermal servo-control system at delivery could prevent heat loss during this delicate phase and increase the percentage of very low birth weight infants (VLBWI) in the normal thermal range (temperature 36.5-37.5°C) at NICU admission. The aim of this study will be to compare two modes of thermal management (with and without the use of a thermal servo-controlled system) for preventing heat loss at birth in VLBWI infants.

ELIGIBILITY:
Inclusion Criteria:

1. Estimated birth weight <1500 g and/or gestational age <30+6 weeks (and)
2. Inborn (and)
3. Parental consent

Exclusion Criteria:

1. Major congenital malformations (i.e. cardiac disease, defects of abdominal wall, ...);
2. Outborn;
3. Parental refusal to participate to the study.

Ages: 1 Minute to 1 Minute | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 440 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-02-29 (Actual); Study Completion 2020-02-29 (Actual)

PRIMARY OUTCOMES:
Proportion of neonates in the normal thermal range (temperature 36.5-37.5°C) at NICU admission | 30 minutes

SECONDARY OUTCOMES:
Proportion of neonates with temperature less than 36.0°C at NICU admission | 30 minutes
Proportion of neonates with mild hypothermia (temperature 36.0-36.4°C) at NICU admission | 30 minutes
Proportion of hyperthermic neonates (temperature >38.0°C) at NICU admission | 30 minutes
Temperature at 1 hour after NICU admission | 1 hour
Proportion of ineonates with ntraventricular hemorrhage (grade I-IV) | 7 days
Propoertions of neoantes with respiratory distress syndrome | 3 days
Proportion of neonates with late onset sepsis | 14 days
Proportion of neonates with bronchopulmonary dysplasia | 36 gestational weeks
Proportion of deaths | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Padova, Padua, Italy

REFERENCES:
- [Derived] Cavallin F, Doglioni N, Allodi A, Battajon N, Vedovato S, Capasso L, Gitto E, Laforgia N, Paviotti G, Capretti MG, Gizzi C, Villani PE, Biban P, Pratesi S, Lista G, Ciralli F, Soffiati M, Staffler A, Baraldi E, Trevisanuto D; Servo COntrol for PReterm Infants (SCOPRI) Trial Group. Thermal management with and without servo-controlled system in preterm infants immediately after birth: a multicentre, randomised controlled study. Arch Dis Child Fetal Neonatal Ed. 2021 Nov;106(6):572-577. doi: 10.1136/archdischild-2020-320567. Epub 2021 Feb 17. PMID 33597230